CLINICAL TRIAL: NCT07283692
Title: NEOadjuvant SERplulimab Plus Weekly PaclitaxEl and carboplatiN in Triple-negative Breast Cancer: a Prospective, Single-arm, Multicenter, Phase 2 Clinical Trial
Brief Title: Neoadjuvant Serplulimab Plus Weekly Paclitaxel and Carboplatin in TNBC (Neo-SERPENT)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Wenjin Yin, Deputy Chief of Breast Surgery Department, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY2025-277-A
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Triple Negative Breast Cancer
Keywords: breast cancer; neoadjuvant; serplulimab
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant serplulimab (Experimental): serplulimab in combination with weekly paclitaxel and carboplatin as neoadjuvant therapy
  Interventions: Drug: Serplulimab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Serplulimab — 1.5mg/kg qw, start from C1D15
Drug: Paclitaxel — 80mg/m^2 qw
Drug: Carboplatin — AUC=1.5, D1, 8, 15, every 28 days

SUMMARY:
This is an prospective, open label, multicenter study to evaluate the efficacy and safety of neoadjuvant serplulimab plus weekly paclitaxel and carboplatin in patients with triple-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female, Aged ≥18 and ≤70 years
* Histologically confirmed triple negative breast cancer (ER<10%, PR<10%, and HER2 negative)
* Subjects with at least one evaluable lesion
* ECOG 0-1
* Adequate organ function

Exclusion Criteria:

* Metastatic disease (Stage IV)
* Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test;Female patients of childbearing age that are reluctant to take effective contraceptive measures throughout the trial period

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with pCR | 1-2 weeks after surgery
  Number of patients with pathological complete response/Number of all eligible patients

SECONDARY OUTCOMES:
Proportion of patients with adverse events | From the date of starting neoadjuvant therapy to the end of the treatment (up to approximately 1 year)
  Number of patients with adverse events during neoadjuvant therapy assessed according to the NCI CTCAE v5.0/Number of all eligible patients

CONTACTS AND LOCATIONS:
Overall Officials: Wenjin Yin, M.D., Principal Investigator — Renji Hospital,School of Medicine, Shanghai Jiaotong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided